CLINICAL TRIAL: NCT01889108
Title: Feasibility Study of Supporting Play, Exploration, & Early Development Intervention (SPEEDI) for Infants Born Preterm
Brief Title: Feasibility Study of SPEEDI
Acronym: SPEEDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCU_HM13949
Record Dates: First submitted 2013-06-13; First posted 2013-06-28 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Premature
Keywords: Premature; Development; Motor; Cognitive; Parent
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual care
- Intervention group (Experimental): Intervention with SPEEDI
  Interventions: Behavioral: SPEEDI

INTERVENTIONS:
Behavioral: SPEEDI — Behavior intervention combining parent education and physical therapy intervention for preterm infants
  Other Names: Developed for this study
  Arms: Intervention group

SUMMARY:
The proposed feasibility study will evaluate the investigators ability to conduct a clinical trial of a novel intervention (SPEEDI) which addresses a striking gap in the literature. Supporting Play, Exploration, and Early Development Intervention (SPEEDI) differs from current early intervention practices in 2 important ways. First it bridges the traditional gap in services from the Neonatal Intensive Care Unit (NICU) to home providing ongoing and intensive support for developmental activities when parents are establishing care giving routines. Second, in contrast to wide-ranging intervention provided by current early intervention models, SPEEDI uses an action perception model to target specific behaviors which lead to improved early motor abilities and provide a foundation for learning.[6] The purpose of this feasibility study is to extend the investigators preliminary data and evaluate the feasibility of conducting a randomized control trial to evaluate the efficacy of SPEEDI.

ELIGIBILITY:
Inclusion Criteria:

* infants born preterm at 34 weeks Post Menstrual Age (PMA) or less
* medically stable,
* off ventilator support,
* demonstrate thermoregulation in an open crib by 35 weeks of PMA,
* live within 60 minutes of the hospital, and
* have one parent who is English speaking and willing to participate in the study intervention and assessments

Exclusion Criteria:

* genetic syndrome or
* musculoskeletal deformity

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Test of Infant Motor Performance | Change from baseline to the end of intervention at 3 months of adjusted age
  Assessment of motor development
Problem Solving Behaviors | end of intervention at 3 months of adjusted age
  Early infant problem solving
Reaching | end of intervention at 3 months of adjusted age
  Reaching and object interaction measures

SECONDARY OUTCOMES:
Parent Child Interactions | End of intervention at 3 months of adjusted age
  Behavioral coding of parent child interactions

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States